CLINICAL TRIAL: NCT03531320
Title: Open-Label, Multicenter Study of D07001-Softgel Capsules (Oral Gemcitabine Hydrochloride) in Subjects With Unresectable, Metastatic or Locally Advanced Gastrointestinal (GI) Cancer in Dose-Escalation Phase and in Subjects With Advanced Biliary Tract Cancer (BTC) Following Primary Chemotherapy or Combined Chemoradiotherapy (CCRT) in Dose-Expansion Phase
Brief Title: Study of D07001-Softgel Capsules in Subjects With Gastrointestinal Cancer in Dose-Escalation Phase and in Subjects With Biliary Tract Cancer in Dose-Expansion Phase
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InnoPharmax Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Inno-GO-03
Record Dates: First submitted 2018-04-10; First posted 2018-05-21 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Gastrointestinal Cancer; Biliary Tract Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Intervention Model Description: Part 1 of the study comprises a sequential dose escalation to identify dose-limiting toxicity (DLT) and establish the maximum tolerated dose (MTD), if any, of D07001-softgel in patients with unresectable locally advanced or metastatic GI cancer. Part 1 will follow a 3+3 dose escalation scheme at predefined dose levels. There will be sequential cohorts of 3 to 6 patients each with increasing doses of 40 mg, 60 mg, 80 mg, 120 mg, and 160 mg per cohort.
  In Part 2 of the study, D07001-softgel will be administered at the 2 dose levels selected for expansion from Part 1 of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1:Dose-Escalation Phase (Experimental): 40 mg D07001-softgel capsules 60 mg D07001-softgel capsules 80 mg D07001-softgel capsules 120 mg D07001-softgel capsules 160 mg D07001-softgel capsules
  Interventions: Drug: D07001-softgel capsules
- Part 2: Dose-Expansion Phase (Phase 2) (Experimental): higher dose-expansion of D07001-softgel capsules lower dose-expansion of D07001-softgel capsules
  Interventions: Drug: D07001-softgel capsules

INTERVENTIONS:
Drug: D07001-softgel capsules — Active Ingredient:Gemcitabine hydrochloride

SUMMARY:
Part 1: Dose-Escalation Phase (Phase 1b) The primary objective is to assess the safety and tolerability of increasing doses of D07001 softgel in patients with unresectable locally advanced or metastatic gastrointestinal (GI) cancer.

Part 2: Dose-Expansion Phase (Phase 2) The primary objective is to assess the safety and tolerability of D07001 softgel in patients who have achieved stable disease or better following first line chemotherapy or combined chemoradiotherapy (CCRT) for unresectable metastatic or locally advanced biliary tract cancer (BTC)

DETAILED DESCRIPTION:
This open label, multicenter study will be conducted in 2 parts: a dose-escalation phase (Part 1) and a dose-expansion phase (Part 2).

In both Part 1 and Part 2, eligible patients will be assigned to receive oral D07001-softgel on Days 1, 3, 5, 8, 10, 12, 15, 17, and 19 of a 21-day cycle (9 doses per cycle).

Part 1: Dose Escalation Phase (Phase 1b) Part 1 of the study will follow a 3+3 dose escalation scheme at predefined dose levels. There will be sequential cohorts of 3 to 6 patients each with increasing doses of 40 mg, 60 mg, 80 mg, 120 mg, and 160 mg per cohort. There will be no intra patient dose escalation. Cycle 1 (21 days) is defined as the dose limiting toxicity (DLT) assessment period.

Part 2: Dose Expansion Phase (Phase 2) In Part 2 of the study, eligible patients will be randomized in a 1:1 ratio to receive D07001-softgel in an open label manner at 1 of the 2 dose levels selected for expansion. Twenty (20) patients will be enrolled to each dose expansion cohort. Patients will be treated until withdrawal from treatment due to disease progression according to RECIST v1.1, withdrawn consent, or when another treatment discontinuation criterion is met. Patients who are discontinued from study drug for reasons other than disease progression or toxicity in the first 2 cycles of Part 2 will be replaced.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of a signed and dated written Informed Consent Form (ICF) prior to any study specific procedures
2. Male or female patients aged 18 years or older at screening (aged 20 years or older in Taiwan)
3. Histopathological or cytologic diagnosis of unresectable, metastatic or locally advanced GI cancer (Part 1) or unresectable metastatic or locally advanced BTC (cholangiocarcinoma or gallbladder cancer; Part 2)
4. Part 1 only: Refractory to or have relapsed from all standard therapies of advanced GI malignancy
5. Part 2 only:

   1. Achieved stable disease or better, based on the Investigator's assessment, in response to first line systemic therapy or CCRT, with continued stable disease or better based on imaging studies obtained as part of screening
   2. Completed first line systemic therapy (with 2-8 cycles of chemotherapy with a gemcitabine based regimen) or CCRT, based on the local standard of care and preferences in the participating countries Note: No more than 30% of patients enrolled in Part 2 will have received CCRT
6. No more than 60 days have elapsed between completion of the prior line of chemotherapy or CCRT and enrollment
7. Part 2 only: Patient has not received intervening systemic therapy since first line treatment
8. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-2 in Part 1 and 0-1 in Part 2
9. Life expectancy is >12 weeks
10. Adequate bone marrow function, demonstrated by:

    1. Absolute neutrophil count (ANC) ≥1,500 cell/mm3
    2. Platelet count ≥100,000 cells/mm3
    3. Hemoglobin ≥9 g/dL
11. Adequate liver function, demonstrated by:

    1. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 x upper limit of normal (ULN), or ≤5.0 x ULN in the case of liver metastases
    2. Total bilirubin ≤1.5 x ULN
    3. Albumin ≥3.0 g/dL
    4. International normalized ratio (INR) <1.5
12. Adequate renal function, demonstrated by:

    1. Serum creatinine ≤1.5 x ULN
    2. Creatinine clearance ≥ 60 mL/min calculated by Cockcroft-Gault formula or directly measured with 24 hr urine collection
13. If a woman of childbearing potential, the patient has a negative serum pregnancy test at screening and is not breastfeeding
14. If a woman of childbearing potential, patient must use a medically acceptable form of contraception as 2 barrier methods (e.g., combination of condom, diaphragm, or intrauterine device), hormonal contraception (estrogen or progesterone agents) or 1 barrier method in combination with spermicide. Birth control is required 1 month prior to screening, for the duration of their study participation, and for 1 month after the end of the study; female partners of male patients must adhere to the same birth control methods.
15. Patient is willing to comply with protocol-required visit schedule and visit requirements

Exclusion Criteria:

1. Part 2 only: More than one prior chemotherapy regimen for unresectable metastatic or locally advanced BTC Note: prior radiation (with or without radiosensitizing doses of chemotherapy) or fluoropyrimidine chemotherapy are allowed as postsurgical adjuvant therapy.
2. Part 2 only: Received any systemic therapy (chemotherapy, biologics, immunotherapy, or investigational agents) for metastatic disease other than gemcitabine based chemotherapy or CCRT for locally advanced BTC
3. Diagnosis of active malignancy (other than GI cancer [Part 1] or BTC [Part 2]) within the past 2 years, except nonmelanoma skin carcinoma and carcinoma-in-situ of uterine cervix treated with curative intent
4. Prior discontinuation of gemcitabine because of pulmonary or hepatic toxicity or hemolytic uremic syndrome (HUS) or hypersensitivity, allergic reaction, or intolerance
5. Any GI disorder which would significantly impede absorption of an oral agent
6. Known brain or leptomeningeal metastases
7. Surgery or radiation therapy within the past 28 days
8. Part 2 only: Evidence of disease progression, based on the Investigator's assessment, on the screening computed tomography (CT) scan or magnetic resonance imaging (MRI) scan
9. Any active disease or condition that would not permit compliance with the protocol
10. Residual toxicity from prior chemotherapy or CCRT that is Grade ≥2 (residual Grade 2 neuropathy and alopecia are permitted)
11. Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, unstable angina, congestive heart failure, or New York Heart Association [NYHA] Grade 2 or greater), or uncontrolled serious cardiac arrhythmia
12. Patient has a history of drug or alcohol abuse within last year
13. Patient has documented cerebrovascular disease
14. Patient has a seizure disorder not controlled on medication (based on decision of Investigator)
15. Patient received an investigational agent within 28 days of enrollment
16. Patients with uncontrolled active viral, bacterial, or systemic fungal infection
17. Patient has known human immunodeficiency virus (HIV) infection
18. Patient has hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection in medical history. If positive results are not indicative of true active or chronic infection, the patient can enter the study after discussion and agreement between the Investigator and the Clinical Research Organization (CRO) Medical Monitor
19. Patient has received yellow fever vaccine or other live attenuated vaccine(s) within the 4 weeks prior to screening
20. Patient has any other serious medical condition that, in the Investigator's medical opinion, would preclude safe participation in, and compliance with, a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, Ph. D, Principal Investigator — National Cheng-Kung University Hospital
Locations (4):
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1:Dose-Escalation Phase_40mg: 40 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase_60mg: 60 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase_80mg: 80 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase_120mg: 120 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase_100mg: 100 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
  Due to safety concern, SMC members recommended adding a 100mg dose group instead of the 160mg dose.
Period: Overall Study
Arm/Group | Part 1:Dose-Escalation Phase_40mg | Part 1:Dose-Escalation Phase_60mg | Part 1:Dose-Escalation Phase_80mg | Part 1:Dose-Escalation Phase_120mg | Part 1:Dose-Escalation Phase_100mg
Started | 4 | 3 | 3 | 6 | 3
Completed | 3 | 3 | 3 | 6 | 3
Not Completed | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total 19 subjects
Groups:
- Part 1:Dose-Escalation Phase Level 1: Cohort 1: 40 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase Level 2: Cohort 2: 60 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase Level 3: Cohort 3: 80 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase Level 4: Cohort 4: 120 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase Level 5: Cohort 5: 100 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Total: Total of all reporting groups
Arm/Group | Part 1:Dose-Escalation Phase Level 1 | Part 1:Dose-Escalation Phase Level 2 | Part 1:Dose-Escalation Phase Level 3 | Part 1:Dose-Escalation Phase Level 4 | Part 1:Dose-Escalation Phase Level 5 | Total
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 3 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (13.52) | 57.7 (10.69) | 54.7 (13.01) | 55.5 (10.88) | 55.7 (15.50) | 58.3 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 1 | 1 | 4
  Male | 3 | 3 | 2 | 5 | 2 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 3 | 3 | 6 | 3 | 19
Region of Enrollment [Number; unit: participants]
  Taiwan | 4 | 3 | 3 | 6 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Establish the Maximum Tolerated Dose (MTD)
Description: MTD will be defined based on the number of dose limiting toxicities (DLT) in subjects at each dose level.
  DLT definition: In Part 1 of the study, any of the following AEs occurring during Cycle 1 will be classified as DLTs, if there is a reasonable possibility that it is related to the study drug
  * Hematologic:
    * Grade 4 neutropenia lasting >7 days
    * Febrile neutropenia (defined as neutropenia Grade ≥3 and a body temp ≥38.3°C)
    * Grade ≥3 neutropenic infection
    * Grade 4 anemia
    * Grade ≥3 thrombocytopenia with bleeding
    * Grade 4 thrombocytopenia
  * Non-hematologic:
    o Grade ≥3 toxicities that are considered clinically significant, except those that have not been maximally treated (e.g., nausea, vomiting, diarrhea*) or can be easily treated (e.g., electrolyte abnormalities).
  * Failure to deliver at least 6 of the planned 9 doses during Cycle 1 due to treatment-related toxicities.
  * Upon the second occurrence of a toxicity leading to a dose hold.
Time Frame: During Cycle 1 of treatment (each cycle is 21 days) for each subject
Population: Only Part 1 was conducted. 2 DLTs were happened in 120mg group, so the MTD is 100mg.
Measure: Number; unit: mg
Groups:
- Part 1:Dose-Escalation Phase: 40 mg D07001-softgel capsules 60 mg D07001-softgel capsules 80 mg D07001-softgel capsules 120 mg D07001-softgel capsules 100 mg D07001-softgel capsules (additional cohort)
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
Arm/Group | Part 1:Dose-Escalation Phase
Number analyzed (Participants) | 19
mg | 100

2. Primary Outcome: Part 1 : Incidence of Adverse Events (AEs)/ Serious Adverse Event (SAEs)
Description: AEs will be assessed via the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Time Frame: From date of informed consent to 30-day follow-up visit for each subject, an average of 10 months
Population: Please refer to the Adverse Event tables for specifics.
Measure: Number; unit: participants
Groups:
- Part 1:Dose-Escalation Phase Level 1: 40 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase Level 2: 60 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase Level 3: 80 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase Level 4: 120 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
- Part 1:Dose-Escalation Phase Level 5: 100 mg D07001-softgel capsules
  D07001-softgel capsules: Active Ingredient:Gemcitabine hydrochloride
Arm/Group | Part 1:Dose-Escalation Phase Level 1 | Part 1:Dose-Escalation Phase Level 2 | Part 1:Dose-Escalation Phase Level 3 | Part 1:Dose-Escalation Phase Level 4 | Part 1:Dose-Escalation Phase Level 5
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 3
participants
  Related to study drug SAEs | 0 | 0 | 0 | 2 | 1
  Related to study drug AEs | 2 | 2 | 3 | 6 | 3
  DLTs | 0 | 0 | 0 | 2 | 0

3. Primary Outcome: Part 2: Incidence of Dose Modifications, Including Dose Reduction, Interruption, or Discontinuation of Study Drug
Description: To measure ratio of total subjects who experienced the dose modifications including dose reduction, interruption, or discontinuation of study drug due to AEs.
Time Frame: First dose through last dose for each subject, an average of 8 months
Population: Only Part 1 was conducted.
Arm/Group | Part 2: Dose-Expansion Phase (Phase 2)
Number analyzed (Participants) | 0

4. Secondary Outcome: Part 1: Pharmacokinetics (PK)- Cmax
Description: PK would be analyzed by maximum concentration (Cmax) of dFdC
Time Frame: Cycle 1 Days 1 and 15
Population: Only Part 1 was conducted.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1:Dose-Escalation Phase Level 1 | Part 1:Dose-Escalation Phase Level 2 | Part 1:Dose-Escalation Phase Level 3 | Part 1:Dose-Escalation Phase Level 4 | Part 1:Dose-Escalation Phase Level 5
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 3
ng/mL
  Cycle 1 Day 1 | 13.67 (7.58) | 42.97 (27.14) | 7.37 (5.68) | 37.24 (23.84) | 24.05 (17.43)
  Cycle 1 Day 15 | 14.45 (13.93) | 12.93 (2.84) | 10.66 (9.15) | 18.47 (13.31) | 13.28 (7.92)

5. Secondary Outcome: Part 1: PK- AUC
Description: PK would be analyzed by Area Under Curve (AUC) of dFdC
Time Frame: Cycle 1 Days 1 and 15
Population: Only Part 1 was conducted.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1:Dose-Escalation Phase Level 1 | Part 1:Dose-Escalation Phase Level 2 | Part 1:Dose-Escalation Phase Level 3 | Part 1:Dose-Escalation Phase Level 4 | Part 1:Dose-Escalation Phase Level 5
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 3
h*ng/mL
  Cycle 1 Day 1 | 12.35 (7.12) | 41.14 (4.42) | 11.59 (8.83) | 62.79 (42.10) | 54.40 (44.19)
  Cycle 1 Day 15 | 12.71 (13.07) | 19.50 (3.74) | 14.05 (10.30) | 35.20 (33.29) | 36.96 (31.35)

6. Secondary Outcome: Part 2: Pharmacokinetics (PK)- Cmax
Description: PK would be analyzed by maximum concentration (Cmax) of dFdC
Time Frame: Cycle 1 Days 1, 8, and 15; Cycle 1 Day 15 and Cycle 2 Day 1 for food-effect cohort only
Population: Only Part 1 was conducted.
Arm/Group | Part 2: Dose-Expansion Phase (Phase 2)
Number analyzed (Participants) | 0

7. Secondary Outcome: Part 2: PK- AUC
Description: PK would be analyzed by Area Under Curve (AUC) of dFdC
Time Frame: Cycle 1 Days 1, 8, and 15; Cycle 1 Day 15 and Cycle 2 Day 1 for food-effect cohort only
Population: Only Part 1 was conducted.
Arm/Group | Part 2: Dose-Expansion Phase (Phase 2)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The Adverse event information was collected and assessed in relation to baseline for study patients from the first dose of treatment until 30 days after discontinuation of treatment.
Description: Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 The AEs/SAEs were collected in relation to study drug.
Arm/Group | Part 1:Dose-Escalation Phase Level 1 | Part 1:Dose-Escalation Phase Level 2 | Part 1:Dose-Escalation Phase Level 3 | Part 1:Dose-Escalation Phase Level 4 | Part 1:Dose-Escalation Phase Level 5 | Part 2: Dose-Expansion Phase (Phase 2)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/6 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 2/6 | 1/3 | 0/0
Other Adverse Events (participants affected / at risk) | 2/4 | 2/3 | 3/3 | 6/6 | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:Dose-Escalation Phase Level 1 (N=4) | Part 1:Dose-Escalation Phase Level 2 (N=3) | Part 1:Dose-Escalation Phase Level 3 (N=3) | Part 1:Dose-Escalation Phase Level 4 (N=6) | Part 1:Dose-Escalation Phase Level 5 (N=3) | Part 2: Dose-Expansion Phase (Phase 2) (N=0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0
hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:Dose-Escalation Phase Level 1 (N=4) | Part 1:Dose-Escalation Phase Level 2 (N=3) | Part 1:Dose-Escalation Phase Level 3 (N=3) | Part 1:Dose-Escalation Phase Level 4 (N=6) | Part 1:Dose-Escalation Phase Level 5 (N=3) | Part 2: Dose-Expansion Phase (Phase 2) (N=0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (3) | 3 (7) | 2 (5) | 0
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (9) | 0 (0) | 0
Fever (General disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (3) | 1 (1) | 0
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 0
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0
Faitigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 (2) | 0 | NA
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 (2) | 0 | NA
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 (2) | 0 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between Principal Investigators and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT03531320/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT03531320/SAP_001.pdf